



| Participant name: | | | | |
|---|---|---|---|---|
| Patient Identification Number for this trial: | | | | |
| CONSENT FORM | | | | |
| Title of Project: ObeSity related Colorectal Adenoma Risk: The OSCAR Study | | | | |
| Name of Researcher: <b>Professor Colin Rees</b> Please ini | | | | <b>5</b> S |
| 1. | I confirm that I have read and understand the information sheet dated (version) for the above study. 1. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | ] |
| 3. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected, but information collected up to that point may still be used by the study team. | | | |
| <ul><li>4.</li><li>5.</li></ul> | | | | |
| study may be looked at by individuals from South Tyneside NHS Foundation Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | | J |
| 6. I agree to take part in the above study. | | | | |
| Par | ticipant signature | Participant name | Date | |
| Witness signature (if required) | | Witness name | Date | |
| Researcher signature | | Researcher name | Date | |

When completed: original for medical notes, 1 original or photocopy for the patient, 1 original or photocopy for the site file. Consent form: OSCAR Study

Version: 1.0 Date: 14.07.2017